CLINICAL TRIAL: NCT07226063
Title: A Phase II Study of Maintenance Zanzalintinib and Durvalumab in Patients With Advanced Hepatocellular Cancer After Induction Tremelimumab Plus Durvalumab
Brief Title: Maintenance Zanzalintinib and Durvalumab in Participants With Advanced Hepatocellular Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amit Mahipal (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor-Investigator, Amit Mahipal, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE11225
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Zanzalintinib; Durvalumab
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + zanzalintinib (Experimental): Participants will receive treatment regimen of durvalumab and zanzalintinib. Each treatment cycle is 28 days. Participants will continue to receive treatment until disease progression, death, or other reasons for withdrawal.
  Interventions: Drug: Durvalumab; Drug: Zanzalintinib

INTERVENTIONS:
Drug: Durvalumab — Participants will receive 1500 mg durvalumab through intravenous (IV) administration over a period of 60 minutes on Day 1 of each 28-day cycle.
Drug: Zanzalintinib — Participants will receive 60 mg durvalumab orally on Days 1-28 of each 28-day cycle.

SUMMARY:
This research study is for people who were treated with tremelimumab and durvalumab for advanced liver cancer and who are currently receiving durvalumab. Participants in this study will receive a drug called zanzalintinib. They will also continue receiving durvalumab. Studies have shown that patients with advanced liver cancer who had tremelimumab and durvalumab may benefit from taking zanzalintinib while they are taking durvalumab. Zanzalintinib is an investigational drug. This means it has not been approved by the U.S. Food and Drug Administration (FDA) for the treatment of patients with advanced liver cancer. Durvalumab is approved by the FDA for patients with advanced liver cancer. The purpose of this study is to find out if taking zanzalintinib with durvalumab will improve how long people with advanced liver cancer will live.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) (liver cancer) is the third most common cause of cancer-related deaths in the world. In 2020, there were over 900,000 new HCC cases and about 830,000 deaths. For early stages, surgery and liver transplantation can sometimes cure the disease. However, most people with HCC are diagnosed in later, advanced stages of the disease, where systemic (whole body) treatment is the only option. Even with these systemic treatment options, median overall survival is still less than 2 years. Zanzalintinib is an oral drug that targets kinases, which are proteins that help cancer cells grow. It has been shown to work against HCC cancer cells. Researchers hypothesize that the combination of zanzalintinib and durvalumab may help to increase overall survival for people with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have radiographically or histologically or cytologically confirmed hepatocellular cancer. Participants must have advanced cancer (metastatic or unresectable) requiring systemic therapy.
* Participants must be treated with tremelimumab plus durvalumab and have stable disease or response to therapy. Participants must have received 2 to 5 doses of durvalumab prior to starting treatment on the clinical trial.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of durvalumab in combination with zanzalintinib in participants ≤18 years of age, children are excluded from this study.
* ECOG Performance status 0-2.
* Participants must have normal organ and marrow function as defined below based upon meeting all the following laboratory criteria within 14 days before first dose of study treatment:

  * Absolute neutrophil count ≥ 1,500/mcL 1,500/mcL (without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection)
  * Hemoglobin ≥ 9 g/dL (≥ 90 g/L) without transfusion within 2 weeks prior to screening laboratory sample collection.
  * Platelet count ≥ 75,000/mcL
  * Total bilirubin < 2.0 mg/dL or <2x upper limit of normal (ULN) whichever is higher
  * AST (SGOT) ≤ 5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 5 X institutional upper limit of normal
  * Creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft Gault equation
  * International Normalized Ratio (INR) ≤ 1.7 and/or activated partial thromboplastin time (aPTT) ≤ 1.2 x ULN.
  * Serum albumin at least 2.5g/dL for Child-Pugh A
  * Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine
* Child Pugh Score A 5-6
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* At least one index lesion that is measurable based on RECIST 1.1.
* Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from AEs, including immune-related adverse events (irAEs), related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (eg, physiological replacement of corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ Grade 2 fatigue, ≤ Grade 2 hypomagnesemia, ≤ Grade 2 neuropathy are permitted)
* Sexually active fertile participants and their partners must agree to use highly effective method of contraception during the course of the study and for the following durations after the last dose of zanzalintinib or duvalumab whichever was administered later. An additional contraceptive method, such as a barrier method (eg, condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods.

  * through 186 days after the last dose of zanzalintinib or durvalumab for women of childbearing potential (WOCBP) or through 96 days after the last dose of zanzalintinib or durvalumab for men
* Female participants of childbearing potential must not be pregnant at screening. Female participants are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.

Exclusion Criteria:

* Inability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube.
* Participants receiving any other investigational agents concurrently for cancer treatment.
* Participants with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of solid organ or allogeneic stem cell transplant.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. This includes unstable or deteriorating cardiovascular disorders:

  * Congestive heart failure New York Heart Association Class 3 or 4, class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).
  * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.
  * Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study treatment.
  * Note: Participants with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: Participants who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.
  * Prior history of myocarditis.
  * Gastrointestinal (GI) disorders associated with a high risk of perforation or fistula formation:
  * Tumors invading the GI-tract from external viscera
  * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
  * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and participant is asymptomatic
  * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
  * Known gastric or esophageal varices
  * Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks
* Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.

  * Known infection with acute or chronic hepatitis B or C, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness except for participants meeting all of the following criteria: (1) on stable anti-retroviral therapy; (2) CD4+ T cell count ≥ 200/µL; and (3) an undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation. Note: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider. Following illnesses/conditions are also excluded
  * Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  * Malabsorption syndrome.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Requirement for hemodialysis or peritoneal dialysis
* Prior treatment with tyrosine kinase inhibitors for HCC
* Another malignancy that requires active therapy and in the opinion of the Investigator would interfere with monitoring of radiologic assessments of response to Investigational Product, within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy. Incidentally diagnosed prostate cancer is allowed if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6.
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (prednisone >10 mg daily orally) or immunosuppressive agents. Participants with durvalumab related adverse event can be included in the trial as long as participants are not requiring prednisone (or equivalent) > 20 mg daily dosing.
* Pregnant or breastfeeding women are excluded from this study because durvalumab and zanzalintinib has the potential for teratogenic effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated on clinical trial. These potential risks may also apply to other agents used in this study.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors ) and platelet inhibitors (eg, clopidogrel). Note: Participants must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer. Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in participants without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
* Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Note: Participants with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following Principal Investigator approval. Participants with involvement of portal vein or hepatic vessels are allowed to participate.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment.

  * Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Any active, known, or suspected autoimmune disease. Note: Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Known positive test for tuberculosis infection if supported by clinical or radiographic evidence of disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Free thyroxine (FT4) outside the laboratory normal reference range. Asymptomatic participants with FT4 abnormalities can be eligible after Principal Investigator approval.
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.
* Documented hepatic encephalopathy (HE) within 6 months before first dose of study treatment.
* Clinically meaningful ascites (ie, ascites requiring repeated paracentesis) within 6 months before first dose of study treatment.
* Participants who have received any local anticancer therapy including surgery, PEI, RFA, MWA, trans arterial chemoembolization (TACE), or trans arterial radioembolization (TARE) within 28 days prior to first dose of study treatment. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (ie nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) at 16 weeks | Week 16
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR is the percentage of participants whose cancer got better after treatment (i.e. the percentage of participants who had CR or PR, as defined below), and this will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
  Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of one or more new lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Safety and tolerability, as measured by incidence and severity of adverse events | Up to 2 years
  Adverse events will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5. Adverse events will be assessed throughout treatment and up to 30 days after treatment discontinuation for any reason (up to 2 years total).
Overall Survival (OS) | Until death, up to 2 years
  Overall survival (OS) is defined as the duration of time from start of treatment to time of death from any cause.
Clinical benefit rate | Up to 2 years
  Clinical benefit rate is defined as the proportion of participants with objective responses or stable disease (SD), as defined below.
  ORR is the percentage of participants whose cancer got better after treatment (i.e. the percentage of participants who had CR or PR), and this will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of one or more new lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Progression-Free Survival (PFS) | Up to 2 years
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mahipal, MD, MBBS, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No